CLINICAL TRIAL: NCT03769350
Title: Smartphone Cognitive Behavioral Therapy for Major Depressive Disorder: A Randomized, Waitlist-control Trial
Brief Title: Waitlist-Control Trial of Smartphone CBT for Major Depressive Disorder (MDD), Withdrawn
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study must be registered under the sponsor instead of the site, so we have created a new posting in the sponsor's account.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Telefónica S.A. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001670-A
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Smartphone-delivered CBT for MDD (Experimental): 8-week Smartphone delivered CBT for MDD.
  Interventions: Device: Smartphone-delivered CBT for MDD
- 8 Week Waitlist Control (Other): 8-week waitlist control. (Note: participants will be crossed over to 8-week Smartphone-delivered CBT for MDD following the 8-week waitlist control).
  Interventions: Device: Smartphone-delivered CBT for MDD

INTERVENTIONS:
Device: Smartphone-delivered CBT for MDD — 8-week Smartphone-delivered CBT for MDD. In-person cognitive-behavioral therapy (CBT) is an empirically supported treatment for MDD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral activation, and perceptual retraining/mindfulness skills.

SUMMARY:
The investigators are testing the efficacy of Smartphone-delivered cognitive behavioral therapy (CBT) treatment for major depressive disorder (MDD). The investigators hypothesize that participants receiving app-CBT will have greater improvement in QIDS-C scores than those in the waitlist condition at treatment endpoint (week 8).

DETAILED DESCRIPTION:
The primary aims of this study are to test the efficacy of a Smartphone-based CBT treatment for adults with MDD recruited nationally. Eligible subjects (N=112) will be randomly assigned to 8 weeks of Smartphone-delivered CBT for MDD either immediately, or after a 8-week long waiting period (50-50 chance). The investigators hypothesize that Smartphone-delivered CBT for MDD will be feasible and acceptable to individuals with MDD, and that it will lead to greater reductions in MDD symptom severity compared to the passage of time (waitlist control).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current diagnosis of primary DSM-5 MDD, based on MINI
* Currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment (Participants taking psychotropic medication must have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period)
* Past participation in ≥ 4 sessions of CBT for depression
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation as indicated by clinical judgment and/or a score ≥ 2 on the suicidal ideation subscale of the C-SSRS
* Concurrent psychological treatment
* Does not own a supported mobile Smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in MDD severity (QIDS-C) at the end of treatment/waitlist period. | Endpoint (week 8)
  The Quick Inventory of Depressive Symptomatology- Clinician version (QIDS-C) is a clinician-administered interview that assesses depressive symptom severity in the past seven days. It contains 16 items ranging from 0-3, which are summed to generate a total score of depressive symptom severity (range=0-27).

SECONDARY OUTCOMES:
Difference in functional impairment at the end of treatment/waitlist period | Endpoint (week 8)
  Participants who receive app-CBT will have greater improvement on functional impairment (SDS). The SDS uses a Likert scale from 0 (not at all) to 10 (extremely) to assess impairment in occupational, social, and family domains. Higher scores indicate greater impairment.
Difference in quality of life at the end of treatment/waitlist period | Endpoint (week 8)
  Participants who receive app-CBT will have greater improvement on quality of life, assessed using The Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (Q-LES-Q). The Q-LES-Q-SF is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100, with higher scores indicating greater quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States